CLINICAL TRIAL: NCT03507114
Title: An Internet-delivered Rumination Focus Cognitive Behavior Therapy in Romania
Brief Title: Rumination Focus Cognitive Behavior Therapy
Acronym: iRFCBT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: West University of Timisoara (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WUTimisoara-iRFCBT
Record Dates: First submitted 2018-04-19; First posted 2018-04-24 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-02

CONDITIONS: Depression; Dysthymic Disorder; Panic Disorder; Social Phobia; Generalized Anxiety Disorder
Keywords: Rumination; Cognitive behavioural therapy (CBT); Depression; Anxiety
MeSH Terms: conditions — Depression; Dysthymic Disorder; Panic Disorder; Phobia, Social; Generalized Anxiety Disorder; Rumination Syndrome; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Folow-up interviews will be carried out by a different team of assessors (blinded to the treatment condition)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rumination-Focused CBT (RFCBT) (Experimental): RFCBT seeks to change the process of thinking as opposed to the content of thoughts as in standard CBT. The underlying idea is that shifting individuals repetitive negative thinking into the concrete mode will reduce unconstructive ruminations and worries.
  Interventions: Behavioral: Rumination-Focused CBT (RFCBT)
- Wait List Control Group (No Intervention): This arm represents the wait-list comparison group.

INTERVENTIONS:
Behavioral: Rumination-Focused CBT (RFCBT) — RFCBT consists of six online modules that include psycho-education, mood diaries, on-line experiential exercises using audio-recordings & vignettes of participants experiences of the therapy.
  Arms: Rumination-Focused CBT (RFCBT)

SUMMARY:
1. To investigate the efficacy and acceptability of a guided internet-delivered transdiagnostic intervention targeting repetitive negative thinking for individuals with elevated levels of depression and generalized anxiety disorder (mild to moderate clinical symptoms) vs a wait-list control group (WLCG).
2. To investigate the hypothesized mechanism of change: Repetitive negative thinking is reduced first, and consequently the clinical symptoms (depression and/or anxiety) decrease.

DETAILED DESCRIPTION:
The effectiveness of a Rumination Focused Cognitive-Behavioral Treatment (RF-CBT) will be compared with a wait list control group using a randomized control trial (RCT) design in a culture where this has not been tested before. The treatment approach was design to specifically target repetitive negative thinking (e.g., rumination and worries). Specifically, the treatment involves first a functional analysis design to help participants identify when rumination starts, distinguish between helpful versus unhelpful repetitive thinking, and learn more functional responses, and experiential and imagery exercises design to help them shift their thought processing towards concreteness, absorption and compassion. The main goal of the study is to test the effectiveness of this transdiagnostic approach in reducing symptom of depression and anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. be fluent in Romanian,
2. be at least 18 years of age,
3. display elevated levels of worry and/or rumination (e.g., at least one self-report score above the following cut-offs: Penn State Worry Questionnaire Total score > 50 and/or Rumination Response Scale - Brooding sub-scale ≥ 10)
4. have at least a clinical diagnosis of major depressive disorder/dysthymia, and/or generalized anxiety disorder, and/or social anxiety disorder, and/or panic disorder, or any combination of these conditions on Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID-I)

Exclusion Criteria:

1. suicidal plans,
2. changes in the dosage if psychotropic medication during the last month (if present),
3. have bipolar disorder or psychosis (according to medication status)
4. have an alcohol/substance abuse and/or dependence disorder
5. currently take part in other psychological treatment,
6. obvious obstacle to participation (i.e., no current Internet access, long travel plans during the treatment period etc.);
7. have a primary diagnostic of Post-Traumatic Stress Disorder and/or Obsessive Compulsive Disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-07-30 (Estimated); Study Completion 2019-02-27 (Estimated)

PRIMARY OUTCOMES:
Rumination Response Scale -10 items (RRS10) | Absolute values (average score) of RRS10 subscales (Reflection and Brooding) at 8 weeks (post-intervention)
  The Rumination Response Scale -10 items (RRS10) was designed to measure participant's level of rumination. The scale has two subscale: Reflection (5 items) and Brooding (5 items). The score for each subscale ranges from 5 to 20, while the total score ranges from 10 to 40. Low scores are associated with low levels of rumination, while high scores are associated with high levels of rumination.
Perseverative Thinking Questionnaire (PTQ) | Absolute values (average score) of PTQ at 8 weeks (post-intervention)
  Perseverative Thinking Questionnaire (PTQ) was designed to measure participant's level of rumination. The scale is unidimensional and the total score ranges from 0 to 60. Low scores are associated with low levels of rumination, while high scores are associated with high levels of rumination.
Patient Health Questionnaire 9 (PHQ9) | Absolute values (average score) of PHQ9 at 8 weeks (post-intervention)
  The Patient Health Questionnaire 9 (PHQ9) was designed to measure participant's level of depression. The scale is unidimensional and the total score ranges from 0 to 27. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
Generalized Anxiety Disorder 7 (GAD7) | Absolute values (average score) of GAD7 at 8 weeks (post-intervention)
  Generalized Anxiety Disorder 7 (GAD7) was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score ranges from 0 to 21. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.
Social Phobia Inventory (SPIN) | Absolute values (average score) of SPIN at 8 weeks (post-intervention)
  The SPIN was designed to measure participant's level of social phobia. The scale is unidimensional and the total score ranges from 0 to 68. Low scores are associated with low levels of social phobia, while high scores are associated with high levels of social phobia.
Anxiety Sensitivity Index 16 (ASI16) | Absolute values (average score) of ASI at 8 weeks (post-intervention)
  ASI16 was designed to measure participant's level of anxiety sensitivity. The scale is unidimensional and the total score ranges from 0 to 64. Low scores are associated with low levels of anxiety sensitivity, while high scores are associated with high levels of anxiety sensitivity.

SECONDARY OUTCOMES:
Work and Social Adjustment Scale (WSAS) | Absolute values (average score) of WSAS at 8 weeks (post-intervention)
  Work and Social Adjustment Scale (WSAS) was designed to measure symptom interference. The scale is unidimensional and the total score ranges from 0 to 40. Low scores are associated with higher levels of functioning (less interference of clinical symptoms) while high scores are associated with lower levels of functioning (or high interference of clinical symptoms).
Beck Depression Inventory-II (BDI-II) | Absolute values (average score) of BDI-II at 8 weeks (post-intervention)
  The Beck Depression Inventory-II (BDI-II) was designed to measure participant's level of depression. The scale is unidimensional and the total score ranges from 0 to 63. Low scores are associated with low levels of depression, while high scores are associated with high levels of depression.
Penn State Worry Questionnaire (PSWQ) | Absolute values (average score) of PSWQ at 8 weeks (post-intervention)
  The PSWQ was designed to measure participant's level of generalized anxiety or worry. The scale is unidimensional and the total score ranges from 16 to 80. Low scores are associated with low levels of worry, while high scores are associated with high levels of worry.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Tudor Tulbure, PhD, Study Director — West University of Timisoara
Locations (1):
- West University of Timisoara, Timișoara, Timiș County, Romania

IPD SHARING:
Plan to Share IPD: No
Data will be process only at the group level. No individual data will be shared to third parties.

REFERENCES:
- See also: Project official website — https://www.e-cbt.ro/program/brio